CLINICAL TRIAL: NCT04673487
Title: Comparative Study of Commercially Available Typhoid Point of Care Tests to Benchmark Current and Emerging Tools
Brief Title: Commercial Typhoid Tests Validation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: Foundation for Innovative New Diagnostics (FIND) (Unknown)
Responsible Party: Principal Investigator, Dr. Robert Onsare, Dr, Kenya Medical Research Institute
Other Study IDs: SERU 4076
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples obtained from whole blood samples

INTERVENTIONS:
Diagnostic Test: 1. SD Bioline Salmonella Typhi IgG/IgM Fast test, 2. Typhidot Rapid IgG/IgM combo test, 3. TUBEX TF test, 4.Typhoid IgG/IgM Combo Rapid Test CE, 5. Enterocheck WB test, 6. Test-itTM Typhoid IgM test — Evaluation of 11 different Typhoid Rapid Diagnostic Tests that are commercially available internationally and use Blood culture as standard for comparison
  Other Names: 7. Typhoid IgG/IgM Rapid Test Cassette 8. S.typhi-S.paratyphi "A" Direct Antigen Detection test 9. DiaquickS.typhi IgG/IgM Ab test 10. Diaquick S. typhi/paratyphi Ag cassette test 11. Widal test.

SUMMARY:
The study aims to perform a head to head comparison of 11 typhoid tests currently in the market and simultaneously develop a sample set that can be used in future evaluations of emerging technologies. The central objective is to evaluate different Typhoid Rapid Diagnostic Tests (RDTs) that are commercially available internationally for detecting antigens or antibodies to Salmonella Typhi and use Blood culture as standard for comparison. The end point will be to determine estimates of sensitivity and specificity for each test, with 95% confidence interval, using blood culture as reference.

DETAILED DESCRIPTION:
Typhoid fever is an enteric bacterial infection caused by Salmonella enterica serovar Typhi (Salmonella Typhi; S. Typhi). It is an important infectious disease in low- and middle-income countries with over 10.9 million new cases worldwide and 116.8 thousand death in 2017. South Asia and Sub Saharan Africa are the most affected areas of the world. Typhoid fever is common in areas with inadequate sanitation and hygiene. In routine practice, diagnosis of typhoid fever is rarely confirmed as diagnostic tests are unavailable or have limited diagnostic accuracy. Blood culture is the commonest reference standard test but has a lower sensitivity. Alternatives to those methods exist but their performance is poor. The Widal test is still used but as it is based on cross-reactive antigens, it lacks sensitivity and specificity. Clinician often use rapid diagnostic tests to diagnose typhoid. A number of typhoid fever RDTs are commercially available but performance data are not available or not consistent from a study to another. This prospective, multicentre, cross-sectional study will be carried out in 3 hospitals of Nairobi, Kenya. 2000 clinically suspected typhoid cases will be enrolled in this study, blood culture as well as serum for RDT will be received. All typhoid positive and equal typhoid negative serum will be tested for investigational RDTs.

This collaborative study between Kenya Medical Research Institute (KEMRI) and Foundation for Innovative New Diagnostics (FIND) will systematically compare different point of care typhoid tests currently available in the market against the same set of reference standard. The knowledge gained from this trial may benefit health providers' by providing information on diagnostic accuracy of current typhoid test and to decide on utility of these commercial tests. The result obtained from this trial will also be made available to help inform Ministry of Health in Kenya and the World Health Organization (WHO) Essential Diagnostic list (EDL) and stakeholder decision making more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 8 years of age to 65 years of age
* History of fever or axillary temperature of >37.5 °C for at least 3 consecutive days within the last 7 days prior to enrollment
* Clinical suspicion of enteric fever
* One of the following scenarios:

  * Presents to outpatient department or Emergency Department
  * Admitted to hospital within last 12 hours
* Able and willing to provide informed consent (and assent when required)

Exclusion Criteria:

* Unwillingness to participate in the study

  * Inability to provide the required volume of blood
  * Unwillingness to provide blood
  * Known non-infectious / Non typhoid Infectious causes of fever or other alternate diagnosis of fever

Ages: 8 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The trial population will be composed of adults and children suspected of typhoid between 8-65 years of age. Participants will be recruited in 3 hospitals in Nairobi, Kenya.The three hospitals are in Nairobi County and include Mbagathi County Hospital, Mbagathi Road; Medical Missionaries of Mary, Reuben Centre Hospital in Mukuru Slum, Embakasi and City Council Clinic in Mukuru Slum, Embakasi.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity for each test, with 95% confidence interval, using blood culture as reference standard. | At the end of the 6-month sampling period
  Evaluation of different Rapid Diagnostic Tests (RDTs) that are commercially available internationally for detecting antigens or antibodies to Salmonella Typhi and use Blood culture as standard for comparison.

SECONDARY OUTCOMES:
Establishment of a bio repository of well characterized specimen collection at the site available for future assessments of emerging technologies | At the end of the 6-month sampling period
  Establishment of a bio repository of well characterized specimen collection that can be used to evaluate emerging tests.
Estimates of operational characteristics of different RDTs based on quantitative assessment including invalid and indeterminate rates | At the end of the 6-month sampling period
  Evaluation of operational characteristics (invalid and indeterminate rates) of Typhoid RDTs

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Result] Crump JA. Progress in Typhoid Fever Epidemiology. Clin Infect Dis. 2019 Feb 15;68(Suppl 1):S4-S9. doi: 10.1093/cid/ciy846. PMID 30767000
- [Result] Amicizia D, Micale RT, Pennati BM, Zangrillo F, Iovine M, Lecini E, Marchini F, Lai PL, Panatto D. Burden of typhoid fever and cholera: similarities and differences. Prevention strategies for European travelers to endemic/epidemic areas. J Prev Med Hyg. 2019 Dec 20;60(4):E271-E285. doi: 10.15167/2421-4248/jpmh2019.60.4.1333. eCollection 2019 Dec. PMID 31967084
- [Result] Ayukekbong JA, Ntemgwa M, Atabe AN. The threat of antimicrobial resistance in developing countries: causes and control strategies. Antimicrob Resist Infect Control. 2017 May 15;6:47. doi: 10.1186/s13756-017-0208-x. eCollection 2017. PMID 28515903
- [Result] Hamaguchi S, Cuong NC, Tra DT, Doan YH, Shimizu K, Tuan NQ, Yoshida LM, Mai LQ, Duc-Anh D, Ando S, Arikawa J, Parry CM, Ariyoshi K, Thuy PT. Clinical and Epidemiological Characteristics of Scrub Typhus and Murine Typhus among Hospitalized Patients with Acute Undifferentiated Fever in Northern Vietnam. Am J Trop Med Hyg. 2015 May;92(5):972-978. doi: 10.4269/ajtmh.14-0806. Epub 2015 Mar 16. PMID 25778504
- [Result] Moore CE, Pan-Ngum W, Wijedoru LPM, Sona S, Nga TVT, Duy PT, Vinh PV, Chheng K, Kumar V, Emary K, Carter M, White L, Baker S, Day NPJ, Parry CM. Evaluation of the diagnostic accuracy of a typhoid IgM flow assay for the diagnosis of typhoid fever in Cambodian children using a Bayesian latent class model assuming an imperfect gold standard. Am J Trop Med Hyg. 2014 Jan;90(1):114-120. doi: 10.4269/ajtmh.13-0384. Epub 2013 Nov 11. PMID 24218407
- [Result] Baker S, Favorov M, Dougan G. Searching for the elusive typhoid diagnostic. BMC Infect Dis. 2010 Mar 5;10:45. doi: 10.1186/1471-2334-10-45. PMID 20205702
- [Result] Bhaskaran D, Chadha SS, Sarin S, Sen R, Arafah S, Dittrich S. Diagnostic tools used in the evaluation of acute febrile illness in South India: a scoping review. BMC Infect Dis. 2019 Nov 13;19(1):970. doi: 10.1186/s12879-019-4589-8. PMID 31722678
- [Result] Wijedoru L, Mallett S, Parry CM. Rapid diagnostic tests for typhoid and paratyphoid (enteric) fever. Cochrane Database Syst Rev. 2017 May 26;5(5):CD008892. doi: 10.1002/14651858.CD008892.pub2. PMID 28545155
- [Result] Mather RG, Hopkins H, Parry CM, Dittrich S. Redefining typhoid diagnosis: what would an improved test need to look like? BMJ Glob Health. 2019 Oct 31;4(5):e001831. doi: 10.1136/bmjgh-2019-001831. eCollection 2019. PMID 31749999
- [Result] Lim C, Wannapinij P, White L, Day NP, Cooper BS, Peacock SJ, Limmathurotsakul D. Using a web-based application to define the accuracy of diagnostic tests when the gold standard is imperfect. PLoS One. 2013 Nov 12;8(11):e79489. doi: 10.1371/journal.pone.0079489. eCollection 2013. PMID 24265775
- [Result] Lalremruata R, Chadha S, Bhalla P. Retrospective audit of the widal test for diagnosis of typhoid Fever in pediatric patients in an endemic region. J Clin Diagn Res. 2014 May;8(5):DC22-5. doi: 10.7860/JCDR/2014/7819.4373. Epub 2014 May 15. PMID 24995178
- [Result] Begg CB. Statistical methods in medical diagnosis. Crit Rev Med Inform. 1986;1(1):1-22. PMID 3331577
- [Result] Njuguna HN, Cosmas L, Williamson J, Nyachieo D, Olack B, Ochieng JB, Wamola N, Oundo JO, Feikin DR, Mintz ED, Breiman RF. Use of population-based surveillance to define the high incidence of shigellosis in an urban slum in Nairobi, Kenya. PLoS One. 2013;8(3):e58437. doi: 10.1371/journal.pone.0058437. Epub 2013 Mar 7. PMID 23505506
- [Result] Maude RR, de Jong HK, Wijedoru L, Fukushima M, Ghose A, Samad R, Hossain MA, Karim MR, Faiz MA, Parry CM; CMCH Typhoid Study Group. The diagnostic accuracy of three rapid diagnostic tests for typhoid fever at Chittagong Medical College Hospital, Chittagong, Bangladesh. Trop Med Int Health. 2015 Oct;20(10):1376-84. doi: 10.1111/tmi.12559. Epub 2015 Jul 15. PMID 26094960

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04673487/Prot_SAP_ICF_000.pdf